CLINICAL TRIAL: NCT00892957
Title: Clinical Evaluation of Efficacy and Safety of FS VH S/D 500 S-apr for Hemostasis in Subjects Undergoing Vascular Surgery
Brief Title: FS VH S/D 500 S-apr in Vascular Surgery
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Baxter Healthcare Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 550801
Record Dates: First submitted 2009-05-04; First posted 2009-05-05 (Estimated); Results first posted 2012-11-27 (Estimated); Last update posted 2012-11-27 (Estimated); Status verified 2012-10

CONDITIONS: Hemostasis in Participants Receiving Peripheral Vascular Expanded Polytetrafluoroethylene (ePTFE) Graft Prostheses
Keywords: Vascular Surgery; Arterio-arterial bypasses; Arterio-venous (AV) shunts
MeSH Terms: interventions — Fibrin Tissue Adhesive; Solvents; Thrombin; Low Density Lipoprotein Receptor-Related Protein-1

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- FS VH S/D 500 s-apr (Experimental): FS VH S/D 500 s-apr will be applied to the study suture line.
  Interventions: Biological: Fibrin Sealant, Vapor Heated, Solvent/Detergent-treated with 500 IU/ml thrombin and synthetic aprotinin (FS VH S/D 500 s-apr)
- Manual compression with surgical gauze pads (Active Comparator): Dry gauze pads will be positioned to cover the complete study suture line.
  Interventions: Other: Surgical gauze pads

INTERVENTIONS:
Biological: Fibrin Sealant, Vapor Heated, Solvent/Detergent-treated with 500 IU/ml thrombin and synthetic aprotinin (FS VH S/D 500 s-apr) — The actual dose of FS VH S/D 500 s-apr will depend on the length of the suture line and the intensity of bleeding (but shall not exceed 4 mL FS VH S/D 500 s-apr).
  Other Names: Biological two-component fibrin sealant
  Arms: FS VH S/D 500 s-apr
Other: Surgical gauze pads — Manual compression with surgical gauze pads
  Arms: Manual compression with surgical gauze pads

SUMMARY:
The purpose of this study was to compare safety and efficacy of FS VH S/D 500 s-apr (FS) versus manual compression in prosthetic expanded polytetrafluoroethylene (ePTFE) graft placement.

ELIGIBILITY:
Inclusion Criteria:

Preoperative inclusion criteria:

* Subjects undergoing vascular surgery (ie, conduit placement with an ePTFE graft), including arterio-arterial bypasses, including:

  * axillo-femoral
  * axillo-bifemoral
  * aorto-bifemoral
  * ilio-femoral
  * femoro-femoral
  * ilio-popliteal
  * femoro-popliteal (including below knee)
  * femoro-tibial vessel bypass
  * arterio-venous shunting for dialysis access in the upper or lower extremity
* Signed informed consent
* Subject is of childbearing potential, presents with a negative serum or urine pregnancy test, and agrees to employ adequate birth control measures for the duration of the study.
* Subject is willing and able to comply with the requirements of the protocol.

Intraoperative inclusion criterion:

* Suture line bleeding eligible for study treatment is present after surgical hemostasis (ie, suturing). (A definition of eligible suture line bleeding is provided in the study protocol.)

Exclusion Criteria:

Preoperative exclusion criteria:

* Other vascular procedures during the same surgical session (stenting and/or endarterectomy of the same artery are allowed)
* Congenital coagulation disorders
* Prior kidney transplantation
* Heparin-induced thrombocytopenia
* Known hypersensitivity to heparin
* Known hypersensitivity to aprotinin or other components of the product
* Known severe congenital or acquired immunodeficiency (eg, HIV infection or long-term treatment with immunosuppressive drugs (eg, organ transplantation patients)
* Prior radiation therapy to the operating field
* Severe local inflammation at the operating field
* Subject is pregnant or lactating at the time of enrollment
* Subject has participated in another clinical study involving an investigational product (IP) or investigational device within 30 days prior to enrollment or is scheduled to participate in another clinical study involving an IP or investigational device during the course of this study
* Subject has previously participated in this study (Protocol No.: 550801), ie, each subject can only be enrolled once.

Intraoperative Exclusion Criteria:

* Major intraoperative complications that require resuscitation or deviation from the planned surgical procedure
* Intraoperative change in planned surgical procedure, which results in subject no longer meeting preoperative inclusion and/or exclusion criteria, (eg, abandonment of ePTFE graft placement)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 176 (Actual)
Dates: Start 2009-07; Primary Completion 2010-10 (Actual); Study Completion 2010-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Isabella Presch, MD, MBA, Study Director — Baxter Innovations GmbH
Locations (22):
- United States (22):
  - Birmingham, Alabama
  - Tucson, Arizona
  - Fresno, California
  - Orange, California
  - Washington D.C., District of Columbia
  - Jacksonville, Florida
  - Melbourne, Florida
  - Fort Wayne, Indiana
  - Lexington, Kentucky
  - Baton Rouge, Louisiana
  - Saginaw, Michigan
  - Southfield, Michigan
  - Hackensack, New Jersey
  - Buffalo, New York
  - The Bronx, New York
  - Dayton, Ohio
  - Pittsburgh, Pennsylvania
  - San Antonio, Texas
  - Salt Lake City, Utah
  - Charlottesville, Virginia
  - Bellevue, Washington
  - Seattle, Washington

REFERENCES:
- [Background] Saha SP, Muluk S, Schenk W 3rd, Dennis JW, Ploder B, Grigorian A, Presch I, Goppelt A. A prospective randomized study comparing fibrin sealant to manual compression for the treatment of anastomotic suture-hole bleeding in expanded polytetrafluoroethylene grafts. J Vasc Surg. 2012 Jul;56(1):134-41. doi: 10.1016/j.jvs.2012.01.009. Epub 2012 May 25. PMID 22633423

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were enrolled at 24 clinical sites in the United States, beginning July 2009 and completing in October 2010
Pre-assignment Details: 176 participants were enrolled. 32 were screen failures. 1 was withdrawn by investigator (study coordinator not available to collect data), 2 participants requested withdrawal, 1 participant died prior to screening and prior to receiving study treatment. Therefore, 140 of the 176 enrolled were randomized.
Groups:
- Control - Manual Compression With Surgical Gauze Pads: Dry gauze pads will be positioned to cover the complete study suture line.
Period: Intraoperative Day 0
Arm/Group | FS VH S/D 500 S-apr | Control - Manual Compression With Surgical Gauze Pads
Started | 70 | 70
Completed | 70 | 70
Not Completed | 0 | 0
Period: Postoperative Day 1 Assessment
Arm/Group | FS VH S/D 500 S-apr | Control - Manual Compression With Surgical Gauze Pads
Started | 70 | 70
Completed | 70 | 70
Not Completed | 0 | 0
Period: Between Postoperative Day 1 and Day 14
Arm/Group | FS VH S/D 500 S-apr | Control - Manual Compression With Surgical Gauze Pads
Started | 70 | 70
Completed | 70 | 66
Not Completed | 0 | 4
Not completed — Death | 0 | 2
Not completed — Lost to Follow-up | 0 | 2
Period: Postoperative Day 14 Assessment
Arm/Group | FS VH S/D 500 S-apr | Control - Manual Compression With Surgical Gauze Pads
Started | 68 (Two participants missed postoperative Day 14 assessment, both returned for Day 30 postop assessment) | 66
Completed | 68 | 66
Not Completed | 0 | 0
Period: Postoperative Day 30 Assessment
Arm/Group | FS VH S/D 500 S-apr | Control - Manual Compression With Surgical Gauze Pads
Started | 70 (Two participants missed postoperative Day 14 assessment, both returned for Day 30 postop assessment) | 66
Completed | 70 | 66
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | FS VH S/D 500 S-apr | Control - Manual Compression With Surgical Gauze Pads | Total
Number analyzed (Participants) | 70 | 70 | 140
Age Continuous [Mean (Standard Deviation); unit: years] | 62.5 (12.6) | 66.3 (11.5) | 64.4 (12.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40 | 33 | 73
  Male | 30 | 37 | 67
Region of Enrollment [Number; unit: participants]
  United States | 70 | 70 | 140

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Achieved Hemostasis at 4 Minutes Post Treatment Application.
Description: Hemostasis at the study suture line must be maintained until closure of the surgical wound.
Time Frame: 4 minutes post start of treatment application
Population: Intent to Treat
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- FS VH S/D 500 S-apr: FS VH S/D 500 s-apr was applied to the study suture line
- Control - Manual Compression With Surgical Gauze: Dry gauze pads were positioned to cover the complete study suture line
Arm/Group | FS VH S/D 500 S-apr | Control - Manual Compression With Surgical Gauze
Number analyzed (Participants) | 70 | 70
Percentage of participants | 62.9 [51.2 to 73.6] | 31.4 [21.4 to 42.8]
Statistical Analysis 1: Comparison: FS VH S/D 500 S-apr vs Control - Manual Compression With Surgical Gauze; Test type: Superiority or Other; p < 0.0001, Likelihood ratio chi-square test

2. Secondary Outcome: Percentage of Participants Who Achieved Hemostasis at 6 Minutes Post Treatment Application
Description: Hemostasis at the study suture line must be maintained until closure of the surgical wound.
Time Frame: 6 minutes post start of treatment application
Population: Intent to treat
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | FS VH S/D 500 S-apr | Control - Manual Compression With Surgical Gauze
Number analyzed (Participants) | 70 | 70
percentage of participants | 71.4 [60.2 to 81.1] | 42.9 [31.7 to 54.6]
Statistical Analysis 1: Comparison: FS VH S/D 500 S-apr vs Control - Manual Compression With Surgical Gauze; Test type: Superiority or Other; p = 0.001, Likelihood ratio chi-square test

3. Secondary Outcome: Percentage of Participants Who Achieved Hemostasis at 10 Minutes Post Treatment Application
Description: Hemostasis at the study suture line must be maintained until closure of the surgical wound.
Time Frame: 10 minutes post start of treatment application
Population: Intent to treat
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | FS VH S/D 500 S-apr | Control - Manual Compression With Surgical Gauze
Number analyzed (Participants) | 70 | 70
percentage of participants | 75.7 [64.9 to 84.7] | 55.7 [44.0 to 67.0]
Statistical Analysis 1: Comparison: FS VH S/D 500 S-apr vs Control - Manual Compression With Surgical Gauze; Test type: Superiority or Other; p = 0.012, Likelihood ratio chi-square test

4. Secondary Outcome: Percentage of Participants With Intraoperative Rebleeding After Hemostasis at Study Suture Line
Description: Intraoperative rebleeding at the study suture line after occurrence of hemostasis.
Time Frame: Intraoperative day 0
Population: Intent to treat
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | FS VH S/D 500 S-apr | Control - Manual Compression With Surgical Gauze
Number analyzed (Participants) | 70 | 70
percentage of participants | 5.7 [1.8 to 12.8] | 1.4 [0.1 to 6.1]
Statistical Analysis 1: Comparison: FS VH S/D 500 S-apr vs Control - Manual Compression With Surgical Gauze; Test type: Superiority or Other; p = 0.158, Likelihood ratio chi-square test

5. Secondary Outcome: Percentage of Participants With Postoperative Rebleeding
Description: Any rebleeding requiring surgical re-exploration
Time Frame: Postoperative through day 30 ± 5
Population: Intent to treat
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | FS VH S/D 500 S-apr | Control - Manual Compression With Surgical Gauze
Number analyzed (Participants) | 70 | 70
percentage of participants | 0 [0.0 to 5.1] | 0 [0.0 to 5.1]

6. Secondary Outcome: Percentage of Participants With Graft Occlusion
Description: Determined clinically and defined as absence of blood flow through the graft.
Time Frame: post-op discharge/day 1, post-op day 14 and day 30
Population: Safety Analysis Set
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | FS VH S/D 500 S-apr | Control - Manual Compression With Surgical Gauze
Number analyzed (Participants) | 70 | 70
percentage of participants | 7.1 [2.6 to 14.7] | 11.4 [5.4 to 20.2]
Statistical Analysis 1: Comparison: FS VH S/D 500 S-apr vs Control - Manual Compression With Surgical Gauze; Test type: Superiority or Other; p = 0.380, Likelihood ratio chi-square test

7. Secondary Outcome: Percentage of Participants With Infection at the Surgical Site
Time Frame: post-op discharge/day 1, post-op day 14 and day 30
Population: Safety Analysis Set
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | FS VH S/D 500 S-apr | Control - Manual Compression With Surgical Gauze
Number analyzed (Participants) | 70 | 70
percentage of participants | 10.0 [4.4 to 18.4] | 7.1 [2.6 to 14.7]
Statistical Analysis 1: Comparison: FS VH S/D 500 S-apr vs Control - Manual Compression With Surgical Gauze; Test type: Superiority or Other; p = 0.545, Likelihood ratio chi-square test

8. Secondary Outcome: Number of Participants With Infections by Grade
Description: Infections were recorded according to:
  * Grade I: only dermis affected
  * Grade II: infection invades subcutaneous region but not the arterial implant
  * Grade III: the arterial implant is infected
Time Frame: post-op discharge/day 1, post-op day 14 and day 30
Population: Safety Analysis Set
Measure: Number; unit: participants
Arm/Group | FS VH S/D 500 S-apr | Control - Manual Compression With Surgical Gauze
Number analyzed (Participants) | 70 | 70
participants
  Grade I | 5 | 3
  Grade II | 2 | 1
  Grade III | 0 | 1

9. Secondary Outcome: Vital Signs: Systolic and Diastolic Blood Pressure (BP)- Preoperative Baseline
Time Frame: Within 14 days prior to date of surgery
Population: Safety Analysis Set
Measure: Median (Full Range); unit: mm Hg
Arm/Group | FS VH S/D 500 S-apr | Control - Manual Compression With Surgical Gauze
Number analyzed (Participants) | 70 | 70
mm Hg
  Systolic blood pressure | 139.5 [86 to 197] | 143.5 [90 to 215]
  Diastolic blood pressure | 73.0 [47 to 104] | 76.5 [50 to 113]

10. Secondary Outcome: Percent Change in Vital Signs: Systolic and Diastolic Blood Pressure
Description: Percent Change in Systolic and Diastolic Blood Pressure (BP) Measured as: Preoperative Baseline - Intraoperative Day 0; Preoperative Baseline - Postoperative Day 1; and Preoperative Baseline - Postoperative Day 14
Time Frame: Within 14 days prior to surgery through postoperative day 14
Population: Safety Analysis Set
Measure: Median (Full Range); unit: percent change
Groups:
- FS VH S/D 500 S-apr: Preop Baseline - Intraoperative Day 0; FS VH S/D 500 S-apr: Preop Baseline - Postoperative Day 1; FS VH S/D 500 S-apr: Preop Baseline - Postoperative Day 14: FS VH S/D 500 s-apr was applied to the study suture line
- Control: Preop Baseline - Intraoperative Day 0; Control: Preop Baseline - Postoperative Day 1; Control: Preop Baseline - Postoperative Day 14: Manual compression with surgical gauze - Dry gauze pads were positioned to cover the complete study suture line
Arm/Group | FS VH S/D 500 S-apr: Preop Baseline - Intraoperative Day 0 | Control: Preop Baseline - Intraoperative Day 0 | FS VH S/D 500 S-apr: Preop Baseline - Postoperative Day 1 | Control: Preop Baseline - Postoperative Day 1 | FS VH S/D 500 S-apr: Preop Baseline - Postoperative Day 14 | Control: Preop Baseline - Postoperative Day 14
Number analyzed (Participants) | 70 | 70 | 70 | 70 | 68 | 65
percent change
  Systolic BP | -15.63 [-52.5 to 44.2] | -12.46 [-52.1 to 74.3] | -8.33 [-45.5 to 34.9] | -7.72 [-40.5 to 52.7] | -2.59 [-40.5 to 35.7] | -2.94 [-39.5 to 68.9]
  Diastolic BP (Control Postoperative Day 14 N=64) | -17.29 [-52.9 to 50.0] | -16.87 [-49.5 to 33.9] | -11.58 [-49.4 to 55.3] | -16.84 [-56.6 to 32.8] | -2.64 [-40.2 to 58.2] | -7.30 [-50.5 to 41.4]

11. Secondary Outcome: Vital Signs: Heart Rate - Preoperative Baseline
Time Frame: Within 14 days prior to date of surgery
Population: Safety Analysis Set
Measure: Median (Full Range); unit: beats per minute
Arm/Group | FS VH S/D 500 S-apr | Control - Manual Compression With Surgical Gauze
Number analyzed (Participants) | 70 | 70
beats per minute | 75.0 [52 to 106] | 75.0 [41 to 105]

12. Secondary Outcome: Percent Change in Vital Signs: Heart Rate
Description: Percent Change in Heart Rate Measured as: Preoperative Baseline - Intraoperative Day 0; Preoperative Baseline - Postoperative Day 1; and Preoperative Baseline - Postoperative Day 14
Time Frame: Within 14 days prior to surgery through postoperative day 14
Population: Safety Analysis Set
Measure: Median (Full Range); unit: percent change
Arm/Group | FS VH S/D 500 S-apr: Preop Baseline - Intraoperative Day 0 | Control: Preop Baseline - Intraoperative Day 0 | FS VH S/D 500 S-apr: Preop Baseline - Postoperative Day 1 | Control: Preop Baseline - Postoperative Day 1 | FS VH S/D 500 S-apr: Preop Baseline - Postoperative Day 14 | Control: Preop Baseline - Postoperative Day 14
Number analyzed (Participants) | 70 | 70 | 70 | 70 | 68 | 65
percent change | -6.27 [-34.2 to 32.4] | -2.12 [-37.5 to 123.8] | 5.44 [-22.9 to 82.8] | 4.84 [-36.5 to 84.0] | 5.63 [-20.0 to 79.3] | 0.00 [-23.8 to 81.7]

13. Secondary Outcome: Vital Signs: Respiratory Rate - Preoperative Baseline
Time Frame: Within 14 days prior to date of surgery
Population: Safety Analysis Set
Measure: Median (Full Range); unit: breaths per minute
Arm/Group | FS VH S/D 500 S-apr | Control - Manual Compression With Surgical Gauze
Number analyzed (Participants) | 65 | 68
breaths per minute | 18.0 [12 to 22] | 18.0 [14 to 24]

14. Secondary Outcome: Percent Change in Vital Signs: Respiratory Rate
Description: Percent Change in Heart Rate Measured as: Preoperative Baseline - Postoperative Day 1; and Preoperative Baseline - Postoperative Day 14
Time Frame: Within 14 days prior to surgery through postoperative day 14
Population: Safety Analysis Set
Measure: Median (Full Range); unit: percent change
Arm/Group | FS VH S/D 500 S-apr: Preop Baseline - Postoperative Day 1 | Control: Preop Baseline - Postoperative Day 1 | FS VH S/D 500 S-apr: Preop Baseline - Postoperative Day 14 | Control: Preop Baseline - Postoperative Day 14
Number analyzed (Participants) | 65 | 68 | 62 | 62
percent change | -10.00 [-40.0 to 66.7] | -9.55 [-40.0 to 42.9] | 0.00 [-40.0 to 55.6] | -6.07 [-40.0 to 50.0]

15. Secondary Outcome: Laboratory Values Over Time: Hemoglobin
Time Frame: Preoperative baseline through postoperative Day 14
Population: Safety Analysis Data Set
Measure: Median (Full Range); unit: g/dL
Groups:
- FS VH S/D 500 S-apr: Baseline; FS VH S/D 500 S-apr: Postoperative Day 14: FS VH S/D 500 s-apr, 120 seconds polymerization
- Control Group: Preoperative Baseline; Control Group: Postoperative Day 14: Manual compression with surgical gauze pads
Arm/Group | FS VH S/D 500 S-apr: Baseline | FS VH S/D 500 S-apr: Postoperative Day 14 | Control Group: Preoperative Baseline | Control Group: Postoperative Day 14
Number analyzed (Participants) | 70 | 55 | 67 | 57
g/dL | 12.10 [9.0 to 15.4] | 11.60 [8.1 to 14.5] | 12.20 [9.0 to 18.4] | 11.80 [8.2 to 15.5]

16. Secondary Outcome: Laboratory Values Over Time: Hematocrit
Time Frame: Preoperative baseline through postoperative Day 14
Population: Safety Analysis Data Set
Measure: Median (Full Range); unit: percentage of red blood cells in blood
Arm/Group | FS VH S/D 500 S-apr: Baseline | FS VH S/D 500 S-apr: Postoperative Day 14 | Control Group: Preoperative Baseline | Control Group: Postoperative Day 14
Number analyzed (Participants) | 70 | 55 | 66 | 57
percentage of red blood cells in blood | 37.0 [28 to 50] | 36.0 [28 to 46] | 38.5 [28 to 58] | 37.0 [24 to 49]

17. Secondary Outcome: Laboratory Values Over Time: Erythrocytes
Time Frame: Preoperative baseline through postoperative Day 14
Population: Safety Analysis Data Set
Measure: Median (Full Range); unit: x10^6/µl
Arm/Group | FS VH S/D 500 S-apr: Baseline | FS VH S/D 500 S-apr: Postoperative Day 14 | Control Group: Preoperative Baseline | Control Group: Postoperative Day 14
Number analyzed (Participants) | 70 | 55 | 67 | 57
x10^6/µl | 4.20 [3.1 to 5.3] | 3.90 [2.9 to 5.0] | 4.10 [2.9 to 5.8] | 3.90 [2.4 to 5.7]

18. Secondary Outcome: Laboratory Values Over Time: Leukocytes, Basophils, Eosinophils, Lymphocytes, Neutrophils, and Monocytes
Time Frame: Preoperative baseline through postoperative Day 14
Population: Safety Analysis Data Set
Measure: Median (Full Range); unit: x10^3/µl
Arm/Group | FS VH S/D 500 S-apr: Baseline | FS VH S/D 500 S-apr: Postoperative Day 14 | Control Group: Preoperative Baseline | Control Group: Postoperative Day 14
Number analyzed (Participants) | 70 | 55 | 67 | 57
x10^3/µl
  Leukocytes | 7.105 [2.46 to 14.83] | 8.260 [3.85 to 14.16] | 6.760 [2.93 to 15.00] | 7.980 [3.51 to 13.76]
  Basophils | 0.040 [0.00 to 0.11] | 0.040 [0.00 to 0.11] | 0.040 [0.00 to 0.20] | 0.050 [0.00 to 0.16]
  Eosinophils | 0.180 [0.00 to 0.96] | 0.200 [0.00 to 0.81] | 0.160 [0.05 to 0.61] | 0.220 [0.00 to 0.79]
  Lymphocytes | 1.805 [0.16 to 4.55] | 1.800 [0.29 to 3.74] | 1.700 [0.54 to 4.61] | 1.750 [0.69 to 4.27]
  Neutrophils | 4.585 [0.67 to 11.30] | 5.570 [2.50 to 11.04] | 4.560 [1.32 to 12.19] | 5.150 [2.02 to 10.37]
  Monocytes | 0.370 [0.09 to 1.02] | 0.430 [0.12 to 1.17] | 0.400 [0.15 to 0.98] | 0.460 [0.13 to 1.09]

19. Secondary Outcome: Laboratory Values Over Time: Platelets
Time Frame: Preoperative baseline through postoperative Day 14
Population: Safety Analysis Data Set
Measure: Median (Full Range); unit: x10^3/µl
Arm/Group | FS VH S/D 500 S-apr: Baseline | FS VH S/D 500 S-apr: Postoperative Day 14 | Control Group: Preoperative Baseline | Control Group: Postoperative Day 14
Number analyzed (Participants) | 64 | 52 | 67 | 55
x10^3/µl | 227.0 [77 to 562] | 303.0 [92 to 643] | 239.0 [66 to 646] | 283.0 [116 to 661]

20. Secondary Outcome: Laboratory Values Over Time: Creatinine, Bilirubin, and Blood Urea Nitrogen (BUN)
Time Frame: Preoperative baseline through postoperative Day 14
Population: Safety Analysis Data Set
Measure: Median (Full Range); unit: mg/dL
Arm/Group | FS VH S/D 500 S-apr: Baseline | FS VH S/D 500 S-apr: Postoperative Day 14 | Control Group: Preoperative Baseline | Control Group: Postoperative Day 14
Number analyzed (Participants) | 70 | 57 | 69 | 57
mg/dL
  Creatinine | 1.80 [0.6 to 13.1] | 2.20 [0.7 to 11.1] | 2.90 [0.4 to 12.4] | 4.40 [0.5 to 10.0]
  Bilirubin | 0.30 [0.2 to 1.2] | 0.30 [0.2 to 1.2] | 0.30 [0.2 to 1.4] | 0.30 [0.2 to 1.3]
  BUN | 23.0 [6 to 76] | 23.0 [10 to 77] | 22.0 [7 to 111] | 30.0 [6 to 125]

21. Secondary Outcome: Laboratory Values Over Time: Alanine Aminotransferase (ALT)
Time Frame: Preoperative baseline through postoperative Day 14
Population: Safety Analysis Data Set
Measure: Median (Full Range); unit: U/L
Arm/Group | FS VH S/D 500 S-apr: Baseline | FS VH S/D 500 S-apr: Postoperative Day 14 | Control Group: Preoperative Baseline | Control Group: Postoperative Day 14
Number analyzed (Participants) | 69 | 56 | 65 | 57
U/L | 16.0 [4 to 152] | 16.0 [4 to 95] | 14.0 [4 to 69] | 13.0 [4 to 99]

22. Secondary Outcome: Laboratory Values Over Time: Aspartate Aminotransferase (AST)
Time Frame: Preoperative baseline through postoperative Day 14
Population: Safety Analysis Data Set
Measure: Median (Full Range); unit: U/L
Arm/Group | FS VH S/D 500 S-apr: Baseline | FS VH S/D 500 S-apr: Postoperative Day 14 | Control Group: Preoperative Baseline | Control Group: Postoperative Day 14
Number analyzed (Participants) | 58 | 54 | 63 | 56
U/L | 21.0 [9 to 61] | 20.5 [8 to 81] | 19.0 [8 to 92] | 20.0 [10 to 44]

23. Secondary Outcome: Laboratory Values Over Time: Activated Partial Thromboplastin Time (aPTT)
Time Frame: Preoperative baseline through postoperative Day 14
Population: Safety Analysis Data Set
Measure: Median (Full Range); unit: seconds
Arm/Group | FS VH S/D 500 S-apr: Baseline | FS VH S/D 500 S-apr: Postoperative Day 14 | Control Group: Preoperative Baseline | Control Group: Postoperative Day 14
Number analyzed (Participants) | 65 | 52 | 59 | 53
seconds | 24.40 [18.0 to 150.0] | 25.10 [18.0 to 150.0] | 25.20 [18.2 to 150.0] | 25.80 [19.3 to 150.0]

24. Secondary Outcome: Laboratory Values Over Time: International Normalized Ratio(INR)
Time Frame: Preoperative baseline through postoperative Day 14
Population: Safety Analysis Data Set
Measure: Median (Full Range); unit: ratio
Arm/Group | FS VH S/D 500 S-apr: Baseline | FS VH S/D 500 S-apr: Postoperative Day 14 | Control Group: Preoperative Baseline | Control Group: Postoperative Day 14
Number analyzed (Participants) | 66 | 52 | 59 | 53
ratio | 1.00 [0.9 to 3.6] | 1.00 [0.9 to 4.1] | 1.00 [0.9 to 1.5] | 1.00 [0.9 to 4.1]

25. Primary Outcome: Hemostasis at 4 Minutes After Treatment Application at the Suture Line by Bleeding Severity - Moderate Bleeding
Description: Investigators were shown videos of bleeding severities to standardize assessments.
  Moderate bleeding defined as:
  * Either >25% of the suture line bleeds, or
  * ≥5 suture line bleedings were present, if counting of suture line bleedings was possible, or
  * 1 pulsatile suture line bleeding was present.
Time Frame: 4 minutes post start of treatment application
Population: Intent to Treat
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | FS VH S/D 500 S-apr | Control - Manual Compression With Surgical Gauze
Number analyzed (Participants) | 29 | 27
percentage of participants | 75.9 [58.5 to 88.8] | 48.1 [30.1 to 66.5]

26. Primary Outcome: Hemostasis at 4 Minutes After Treatment Application at the Suture Line by Bleeding Severity - Severe Bleeding
Description: Investigators were shown videos of bleeding severities to standardize assessments.
  Severe bleeding defined as:
  * Either >50% of the suture line bleeds, or
  * ≥10 suture line bleedings were present, if counting of suture line bleedings was possible, or
  * >1 pulsatile suture line bleeding was present, or
  * ≥1 spurting suture line bleeding was present.
Time Frame: 4 minutes post start of treatment application
Population: Intent to Treat
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | FS VH S/D 500 S-apr | Control - Manual Compression With Surgical Gauze
Number analyzed (Participants) | 41 | 42
percentage of participants | 53.7 [38.5 to 68.4] | 20.9 [10.7 to 34.6]

ADVERSE EVENTS:
Time Frame: Throughout the study period, 1 year and 3 months. For SAEs: Recovering/resolving SAEs were followed until resolution, medically stabilized, or 30 days after study completion/termination visit, whichever came first.
Arm/Group | FS VH S/D 500 S-apr | Control - Manual Compression With Surgical Gauze Pads
Serious Adverse Events (participants affected / at risk) | 20/70 | 18/70
Other Adverse Events (participants affected / at risk) | 14/70 | 7/70
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | FS VH S/D 500 S-apr (N=70) | Control - Manual Compression With Surgical Gauze Pads (N=70)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Haematemesis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 2 (2) | 0 (0)
Thrombosis in device (General disorders) | 1 (1) | 0 (0)
Appendicitis perforated (Infections and infestations) | 1 (1) | 0 (0)
Staphylococcal sepsis (Infections and infestations) | 1 (1) | 1 (1)
Wound infection staphylococcal (Infections and infestations) | 1 (1) | 0 (0)
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Postoperative wound infection (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Vascular graft occlusion (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Vascular graft thrombosis (Injury, poisoning and procedural complications) | 2 (4) | 2 (2)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Ischaemic neuropathy (Nervous system disorders) | 1 (1) | 1 (1)
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Arterial thrombosis limb (Vascular disorders) | 1 (1) | 0 (0)
Haematoma (Vascular disorders) | 1 (1) | 0 (0)
Steal syndrome (Vascular disorders) | 1 (1) | 0 (0)
Cardio-respiratory arrest (Cardiac disorders) | 0 (0) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Small intestinal perforation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Multi-organ failure (General disorders) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)
Drug toxicity (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Graft thrombosis (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Incision site cellulitis (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
International normalised ratio increased (Investigations) | 0 (0) | 1 (1)
Hypovolaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | FS VH S/D 500 S-apr (N=70) | Control - Manual Compression With Surgical Gauze Pads (N=70)
Oedema peripheral (General disorders) | 7 (8) | 4 (5)
Operative haemorrhage (Injury, poisoning and procedural complications) | 4 (5) | 1 (2)
Hypotension (Vascular disorders) | 4 (5) | 2 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Baxter's agreements with PIs may vary per requirements of the individual PI, but contain common elements. For this study, PIs are restricted from independently publishing results until the earlier of the primary multicenter publication or 1 year after study completion. Baxter requires a review of results communications (e.g., for confidential information) ≥90 days prior to submission or communication. Baxter may request an additional delay of ≤60 days (e.g., for intellectual property protection)